CLINICAL TRIAL: NCT00937365
Title: A Pilot Randomized Controlled Trial for Complementary and Alternative Medicine Treatment of Pregnancy-Related Low Back Pain.
Brief Title: Pregnancy-Related Low Back Pain and Complementary and Alternative Medicine (CAM) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: The ONE Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5033
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Low Back Pain
Keywords: Pregnancy; Pain; Low back pain; Pubic symphysis pain; CAM; Complementary & Alternative Medicine; Exercise; Chiropractic; Spinal manipulation; Adjustments; Neuroemotional technique; Mind body; Mind body therapy; Attachment; Maternal Fetal relationship; Intrauterine attachment; Heart rate variability; VAS; Visual analog scale; Roland Morris Disability Index
MeSH Terms: conditions — Low Back Pain; Pain; Motor Activity | interventions — Exercise; Manipulation, Spinal; Manipulation, Osteopathic; Mind-Body Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise (Active Comparator): Specific strengthening exercises demonstrated to improve pregnancy-related low back pain are taught to participants of this arm. Additionally, each participant will be evaluated and additional exercises will be prescribed relevant to her particular needs. Study participants of this arm are asked to perform the exercises at home at least once a day. Exercise is recorded in a diary. Participants follow the same study visit schedule as the two other arms.
  Interventions: Behavioral: Exercise
- Spinal Manipulation (Experimental): Women randomized to this arm will be evaluated for spinal subluxations and, if appropriate, treated with chiropractic manipulation. Type of manipulation is determined by presentation. Woman may be manipulated with high velocity low amplitude thrust, blocking, activator, or other appropriate means of manipulating.
  Interventions: Procedure: Spinal Manipulation
- Neuroemotional technique (NET) (Experimental): Neuroemotional technique (NET) is a mind-body technique which combines elements of chiropractic medicine, Chinese medicine, and behavioral psychology. Muscle response testing, a form of functional neurology, and visceral somatic reflexes are used to ascertain whether the pain or dysfunction experienced by the participant has an emotional component. If an emotional component is present, it is identified and the original "triggering" occurrence is identified. The participant creates a snapshot of that original occurrence and while she holds that image in her mind spinal levels which innervate the associated organ are adjusted.
  Interventions: Procedure: Neuroemotional Technique (NET)

INTERVENTIONS:
Behavioral: Exercise — Study visits follow the normal prenatal care schedule (once monthly until 28 weeks, twice monthly until 36 weeks, weekly thereafter). Additional study visits may be necessary if the pain is too intense and requires additional visits.
  Other Names: pelvic tilts; stretch; strengthen; glut squeeze
  Arms: Exercise
Procedure: Spinal Manipulation — Study visits follow the normal prenatal care schedule (once monthly until 28 weeks, twice monthly until 36 weeks, weekly thereafter). Additional study visits may be necessary if the pain is too intense and requires additional visits.
  Other Names: SMT; CMT; chiropractic manipulative therapy; OMT; osteopathic manipulative therapy; adjustment
  Arms: Spinal Manipulation
Procedure: Neuroemotional Technique (NET) — Study visits follow the normal prenatal care schedule (once monthly until 28 weeks, twice monthly until 36 weeks, weekly thereafter). Additional study visits may be necessary if the pain is too intense and requires additional visits.
  Other Names: NET; Mind-body therapy
  Arms: Neuroemotional technique (NET)

SUMMARY:
This study compares three treatments for low back pain that started during pregnancy. The study hypothesizes that exercise, spinal manipulation, and a mind-body technique called neuroemotional technique (NET) equally affect pain intensity and disability associated with pregnancy-related low back pain. The study also hypothesizes that pain intensity and disability levels do not influence maternal heart rate variability (a measure of stress) and intrauterine attachment (a measure of relationship quality). Ten women will additionally provide blood and salivary oxytocin samples during pregnancy and periodically for three months after birth. These women and their babies will also be videotaped playing for 5 minutes at 2 weeks, 6 weeks, and 3 months postpartum.

DETAILED DESCRIPTION:
Pregnancy-related low back pain is experienced by over half of all pregnant women. In the United States it is thought of as a normal constituent of pregnancy. However, in Europe low back pain associated with pregnancy is treated. In the United States pregnancy-related low back pain is thought to resolve with birth. However about 1/3 of women who experience pregnancy-related low back pain continue to experience back pain for one year postpartum. Those women whose low back pain persists into the postpartum period are more at risk of experiencing comorbidities such as postpartum depression.

In the extrauterine life maternal pain limits a mother's ability to securely attach with her child. Furthermore, interpretation of pain intensity is influenced by the type of attachment the individual has with her parents. Little is known how maternal pain may influence intrauterine attachment. Similarly, heart rate variability is influenced by pain and by spinal manipulation in non-pregnant populations. However, normal non-pregnant patterns of heart rate variability are altered during the second and third trimesters of pregnancy, and little is known about why this happens or what this means.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 20-49 years old
* Pregnant with a singleton
* Low back pain began during pregnancy and has lasted more than one week
* Low back pain is reproducible with palpation

Exclusion Criteria:

* Health conditions such as hypertension, diabetes, cancer, thyroid condition etc.
* Pain radiates below knee
* Cannot read English
* Plans to move away from Portland area during pregnancy
* Not willing to be randomized to one of the three arms of the study

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Index | Last study visit prior to birth

SECONDARY OUTCOMES:
Pain Visual Analog Scale | Last Study Visit Before Birth

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gregory, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Benarroch EE. Pain-autonomic interactions: a selective review. Clin Auton Res. 2001 Dec;11(6):343-9. doi: 10.1007/BF02292765. PMID 11794714
- [Background] Borg-Stein J, Dugan SA, Gruber J. Musculoskeletal aspects of pregnancy. Am J Phys Med Rehabil. 2005 Mar;84(3):180-92. doi: 10.1097/01.phm.0000156970.96219.48. PMID 15725792
- [Background] Brage S, Sandanger I, Nygard JF. Emotional distress as a predictor for low back disability: a prospective 12-year population-based study. Spine (Phila Pa 1976). 2007 Jan 15;32(2):269-74. doi: 10.1097/01.brs.0000251883.20205.26. PMID 17224825
- [Background] Depledge J, McNair PJ, Keal-Smith C, Williams M. Management of symphysis pubis dysfunction during pregnancy using exercise and pelvic support belts. Phys Ther. 2005 Dec;85(12):1290-300. PMID 16305268
- [Background] Dipietro JA, Irizarry RA, Costigan KA, Gurewitsch ED. The psychophysiology of the maternal-fetal relationship. Psychophysiology. 2004 Jul;41(4):510-20. doi: 10.1111/j.1469-8986.2004.00187.x. PMID 15189474
- [Background] Hurwitz EL, Morgenstern H, Kominski GF, Yu F, Chiang LM. A randomized trial of chiropractic and medical care for patients with low back pain: eighteen-month follow-up outcomes from the UCLA low back pain study. Spine (Phila Pa 1976). 2006 Mar 15;31(6):611-21; discussion 622. doi: 10.1097/01.brs.0000202559.41193.b2. PMID 16540862
- [Background] Mogren I. Perceived health, sick leave, psychosocial situation, and sexual life in women with low-back pain and pelvic pain during pregnancy. Acta Obstet Gynecol Scand. 2006;85(6):647-56. doi: 10.1080/00016340600607297. PMID 16752254
- [Background] Padua L, Caliandro P, Aprile I, Pazzaglia C, Padua R, Calistri A, Tonali P. Back pain in pregnancy: 1-year follow-up of untreated cases. Eur Spine J. 2005 Mar;14(2):151-4. doi: 10.1007/s00586-004-0712-6. Epub 2004 May 15. PMID 15759172
- [Background] Gartner JG. Thymic involution with loss of Hassall's corpuscles mimicking thymic dysplasia in a child with transfusion-associated graft-versus-host disease. Pediatr Pathol. 1991 May-Jun;11(3):449-56. doi: 10.3109/15513819109064780. PMID 1866363
- [Background] Stuber KJ, Smith DL. Chiropractic treatment of pregnancy-related low back pain: a systematic review of the evidence. J Manipulative Physiol Ther. 2008 Jul-Aug;31(6):447-54. doi: 10.1016/j.jmpt.2008.06.009. PMID 18722200
- [Background] Wadhwa PD. Psychoneuroendocrine processes in human pregnancy influence fetal development and health. Psychoneuroendocrinology. 2005 Sep;30(8):724-43. doi: 10.1016/j.psyneuen.2005.02.004. Epub 2005 Apr 25. PMID 15919579
- [Derived] Peterson CD, Haas M, Gregory WT. A pilot randomized controlled trial comparing the efficacy of exercise, spinal manipulation, and neuro emotional technique for the treatment of pregnancy-related low back pain. Chiropr Man Therap. 2012 Jun 13;20(1):18. doi: 10.1186/2045-709X-20-18. PMID 22694756